CLINICAL TRIAL: NCT01682733
Title: Endoscopic Gastric Reduction for Weight Management: A Pilot Feasibility Study
Brief Title: Endoscopic Gastric Reduction for Weight Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barham K. Abu Dayyeh, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-003195
Record Dates: First submitted 2012-08-27; First posted 2012-09-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Gastric reduction (volume); BMI 30-40
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botulinum toxin at injection site (Experimental): All subjects will have gastroplasty performed using the Overstitch Endoscopic Suturing System. Botulinum toxin will be injected in every other suture site in half of the randomly patients selected.
  Interventions: Drug: Botulinum toxin; Device: Overstitch Endoscopic Suturing System

INTERVENTIONS:
Drug: Botulinum toxin — In this study, Botulinum toxin will be injected in half of the subjects not as a primary treatment modality for obesity, but to retard the muscular grinding gastric activity arount the suture insertion sites to see if it improves the durability of the gastroplasty.
  Other Names: Botox
Device: Overstitch Endoscopic Suturing System — The gastroplasty will be accomplished by a series of intralumenally placed full thickness interrupted sutures through the gastric wall, using the FDA-approved (510K) endoscopic suturing device, the Overstitch Endoscopic Suturing System.

SUMMARY:
The proposed study is a prospective, pilot study to assess the feasibility of a novel endoscopic suturing system to reduce gastric volume by changing the shape of the stomach for the primary treatment of obesity. The investigators aim to recruit ten subjects with a body mass index between 30-40 for this study. Vertical sutures will be performed using the endoscopic suturing system to deploy 10-17 interrupted full thickness sutures. Botulinum toxin(approximately 30 units) will be injected around the sutures insertion sites in half of the subjects randomly to slow down muscular grinding of the stomach to see if it improves durability of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 30 and 40
* Age >18 and ≤50
* Stable weight for 3 months (within 5% of BMI)
* Normal basic labs (CBC, chemistry profile, creatinine)
* Negative pregnancy test for females >18 or ≤ 50

Exclusion Criteria:

* Diabetes
* Unstable coronary artery disease
* Heart failure
* Cardiac arrhythmia
* Cardiac valvular disease
* Obstructive of interstitial lung disease
* Females of child-bearing age >18 or ≤ 50 who are pregnant or lactating
* Mallampati score of 4
* ASA 3 or above
* Previous gastric surgery
* Ulcer disease
* Gastroparesis,
* > 5 cm Hiatal hernia
* Congenital anomalies of the GI tract
* Currently on or prescribed a medication known to affect weight within 3 months of study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Bariatric Quality of Life (BQL) Questionaire | baseline to 3 months

SECONDARY OUTCOMES:
Change from baseline Three factor Eating Questionnaire (TFEQ-R21) | baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Barham K AbuDayyeh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Foundation, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Abu Dayyeh BK, Acosta A, Camilleri M, Mundi MS, Rajan E, Topazian MD, Gostout CJ. Endoscopic Sleeve Gastroplasty Alters Gastric Physiology and Induces Loss of Body Weight in Obese Individuals. Clin Gastroenterol Hepatol. 2017 Jan;15(1):37-43.e1. doi: 10.1016/j.cgh.2015.12.030. Epub 2015 Dec 31. PMID 26748219